CLINICAL TRIAL: NCT02994524
Title: Intersphincteric Approach to Perianal Fistula With High Risk for Postoperative Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser Mohamed Abdel-samii (Other)
Responsible Party: Sponsor-Investigator, Yasser Mohamed Abdel-samii, Lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06379
Record Dates: First submitted 2016-12-08; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: High Transsphincteric Perianal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transsphincteric perianal fistula (Other): Rerouting technique done in patients with high transsphincteric fistula or with high internal opening.
  Interventions: Procedure: Rerouting technique for transsphincteric perianal fistula

INTERVENTIONS:
Procedure: Rerouting technique for transsphincteric perianal fistula

SUMMARY:
.Rerouting operation takes the advantage of minimal recurrence rate as well as minimal incontinence that is associated with less sphincter division,It is indicated in patients with transsphincteric fistula in whom lay open is expected to be associated with significant incontinence .

DETAILED DESCRIPTION:
Lay open is the classic surgical management for Peri Anal fistula,however division of significant portion of anal sphincter may be divided with postoperative fecal incontinence,Many surgical techniques have been described for sphincter preservation ,But unfortunately associated high recurrence rate.Rerouting operation takes the advantage of minimal recurrence rate as well as minimal incontinence that is associated with less sphincter division,It is indicated in patients with transsphincteric fistula in whom lay open is expected to be associated with significant incontinence .The operation is done in tow stages ,the first is to mobilize the transsphincteric part into the inter sphincteric plane thus converting it to intersphincteric fistula which is then laid open , with division of internal sphincter with preserving external sphincter.

ELIGIBILITY:
Inclusion Criteria:

* High arching transsphincteric fistula
* Transsphincteric fistula with high internal opening
* Transsphincteric fistula with short anal canal.
* Horseshoe perianal fistula fulfilling above criteria.

Exclusion Criteria:

* Transsphincteric fistula.
* Low perianal fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Rerouting technique decrease incidence of fecal incontinice after high transsphincteric perianal fistula surgery . | one year

IPD SHARING:
Plan to Share IPD: Undecided